CLINICAL TRIAL: NCT01424345
Title: A Randomized, Controlled Trial Evaluating the Role of ImmuKnow® in the Management of Immunosuppressants Regarding Opportunistic Infections and Acute Rejection in the Renal Transplant Patient
Brief Title: The Role of ImmuKnow® in the Management of Immunosuppressants in the Renal Transplant Patient
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The PI is relocating to another State/ another hospital
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, SC Jeff Chueh, MD, Primary Surgeon, UNOS, CAMC-WV kidney transplant program, CAMC Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1997050
Record Dates: First submitted 2011-08-24; First posted 2011-08-29 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Kidney Transplant Immunosuppression
Keywords: Kidney Transplantation; Immunosuppression; Immune monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Active Comparator): Dosages of immunosuppressants will be given according to the results of conventional post-transplant lab
  Interventions: Drug: adjustment of the dosages of immunosuppressants
- ImmuKnow Study group (Experimental): The dosages of immunosuppressants will be adjusted according to the results of ImmuKnow and conventional post-transplant lab
  Interventions: Drug: adjustment of immunosuppressant dosages

INTERVENTIONS:
Drug: adjustment of immunosuppressant dosages — adjustment of immunosuppressant dosages according to the results of ImmuKnow results and routine post-transplant lab results
  Arms: ImmuKnow Study group
Drug: adjustment of the dosages of immunosuppressants — adjustment of the dosages of immunosuppressants will be done according to the results of conventional post-transplant follow-up lab
  Arms: control group

SUMMARY:
The purpose of this study is to demonstrate whether there are any outcome benefits of a serial ImmuKnow assays in the management of de novo renal transplant recipients.

DETAILED DESCRIPTION:
Background: The management of renal transplant recipients is challenging in keeping a delicate balance of immunosuppression to avoid either infection (overimmunosuppression), or rejection (under-immunosuppression). Conventional clinical parameters are not adequate enough. ImmuKnow (Cylex Inc, Columbia, MD) is an FDA-cleared assay for the detection of cell mediated immune response in populations undergoing immunosuppressive therapy for organ transplant. There have been limited retrospective studies discussing the effectiveness of the ImmuKnow assay. There is no prospective head-to-head trial showing the benefits of periodic ImmuKnow testing.

Objective: To demonstrate whether there are any outcome benefits of a serial ImmuKnow assays in de novo renal transplant recipients Patients and Methods: A prospective, randomized, pilot, controlled 12-month study to compare the outcomes of 2 cohorts of de novo renal transplant patients will be conducted. The outcomes that will be investigated include a combined infection rate (primary end-point), separate infection rates and episodes, acute rejection rate and episodes, quality of life, graft and patient survivals (all secondary end-points). Biopsy of the transplanted kidney is used to confirm rejection whenever possible. Among the study cohort, the patients' immunosuppressants will be adjusted according to the results of a serial ImmuKnow assay besides using conventional clinical parameters; whereas among the control cohort the patients' immunosuppressants will be adjusted according to conventional clinical parameters.

Expected Results: At the end of this study we will be able to learn whether the study cohort patients have less infection, less acute rejection, better allograft function, better quality of life, and better graft or patient survivals.

ELIGIBILITY:
Inclusion Criteria:

1. De novo kidney transplant patients who are eligible for kidney transplant according to UNOS criteria and agree to participate in the study.
2. Patients of both sex aged between 18 to 80 years.

Exclusion Criteria:

* Any patient with a known immunocompromised disease (e.g. patients with AIDS) or leukocytosis(>15,000u/L)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
the combo-infection rates of the 2 cohorts of renal transplant recipients within the 12-month period after a de novo kidney transplantation | 12 months
  The combo-infection is defined as: If a patient either has new onset culture/or serology/or PCR positive bacterial or viral infections; or moderate neutropenia (absolute netrophile count < 1000/microL) or need GCS-F injection or has fever >38.5 % for longer than 24 hrs then he/she is called to have combo- infection. Percentage of such patients will be compared in Immuknow vs. control group.

SECONDARY OUTCOMES:
Event numbers of infection | 12 months
  1.1 Event numbers of new onset infections;1.2 Episodes of patients with moderate neutropenia (< 1000/microL), 1.3 Episodes of patients needing GCS-F; 1.4. Episodes of fever >38.5 % >= 24 hrs.
Percentage of Infection | 12 months
  2.1 percentages of patients with new onset infections; 2.2 percentages of patients with moderate neutropenia, 2.3 percentages of patients needing GCS-F injection; 2.4 percentages of fever >38.5 >= 24 hrs.
Acute rejection | 12 months
  3.1 Episodes of acute rejection; 3.2 Percentages of Acute Rejection.
Life Quality | 12 months
  4.SF-8 QOL index
Allograft function | 12 months
  5.1 serum creatinine levels 5.2 estimated GFR
Graft Survival | 12 months
  6. Graft survival
Patient Survival | 12 months
  7. Patient survival

CONTACTS AND LOCATIONS:
Overall Officials: S Jeff Chueh, MD PhD, Principal Investigator — CAMC Health System, Charleston, WV; Bashir Sankari, MD, Study Director — CAMC Health System, Charleston, Wv
Locations (1):
- CAMC, Charleston, West Virginia, United States

REFERENCES:
- [Background] Kowalski RJ, Post DR, Mannon RB, Sebastian A, Wright HI, Sigle G, Burdick J, Elmagd KA, Zeevi A, Lopez-Cepero M, Daller JA, Gritsch HA, Reed EF, Jonsson J, Hawkins D, Britz JA. Assessing relative risks of infection and rejection: a meta-analysis using an immune function assay. Transplantation. 2006 Sep 15;82(5):663-8. doi: 10.1097/01.tp.0000234837.02126.70. PMID 16969290
- [Background] Reinsmoen NL, Cornett KM, Kloehn R, Burnette AD, McHugh L, Flewellen BK, Matas A, Savik K. Pretransplant donor-specific and non-specific immune parameters associated with early acute rejection. Transplantation. 2008 Feb 15;85(3):462-70. doi: 10.1097/TP.0b013e3181612ead. PMID 18301338
- [Background] Gautam A, Fischer SA, Yango AF, Gohh RY, Morrissey PE, Monaco AP. Cell mediated immunity (CMI) and post transplant viral infections--role of a functional immune assay to titrate immunosuppression. Int Immunopharmacol. 2006 Dec 20;6(13-14):2023-6. doi: 10.1016/j.intimp.2006.09.023. Epub 2006 Oct 24. PMID 17161357
- [Background] Batal I, Zeevi A, Heider A, Girnita A, Basu A, Tan H, Shapiro R, Randhawa P. Measurements of global cell-mediated immunity in renal transplant recipients with BK virus reactivation. Am J Clin Pathol. 2008 Apr;129(4):587-91. doi: 10.1309/23YGPB1E758ECCFP. PMID 18343786
- [Background] Sanchez-Velasco P, Rodrigo E, Valero R, Ruiz JC, Fernandez-Fresnedo G, Lopez-Hoyos M, Pinera C, Palomar R, Leyva-Cobian F, Arias M. Intracellular ATP concentrations of CD4 cells in kidney transplant patients with and without infection. Clin Transplant. 2008 Jan-Feb;22(1):55-60. doi: 10.1111/j.1399-0012.2007.00744.x. PMID 18217906
- [Background] Kowalski R, Post D, Schneider MC, Britz J, Thomas J, Deierhoi M, Lobashevsky A, Redfield R, Schweitzer E, Heredia A, Reardon E, Davis C, Bentlejewski C, Fung J, Shapiro R, Zeevi A. Immune cell function testing: an adjunct to therapeutic drug monitoring in transplant patient management. Clin Transplant. 2003 Apr;17(2):77-88. doi: 10.1034/j.1399-0012.2003.00013.x. PMID 12709071
- [Background] Kobashigawa JA, Kiyosaki KK, Patel JK, Kittleson MM, Kubak BM, Davis SN, Kawano MA, Ardehali AA. Benefit of immune monitoring in heart transplant patients using ATP production in activated lymphocytes. J Heart Lung Transplant. 2010 May;29(5):504-8. doi: 10.1016/j.healun.2009.12.015. Epub 2010 Feb 4. PMID 20133166
- [Background] Huskey J, Gralla J, Wiseman AC. Single time point immune function assay (ImmuKnow) testing does not aid in the prediction of future opportunistic infections or acute rejection. Clin J Am Soc Nephrol. 2011 Feb;6(2):423-9. doi: 10.2215/CJN.04210510. Epub 2010 Nov 18. PMID 21088287
- [Background] Knight RJ, Kerman RH, McKissick E, Lawless A, Podder H, Katz S, Van Buren CT, Kahan BD. Selective corticosteroid and calcineurin-inhibitor withdrawal after pancreas-kidney transplantation utilizing thymoglobulin induction and sirolimus maintenance therapy. Clin Transplant. 2008 Sep-Oct;22(5):645-50. doi: 10.1111/j.1399-0012.2008.00839.x. Epub 2008 Jul 24. PMID 18657156
- [Background] John Ware, Jr, Ph.D., Mark Kosinski, M.A., James E. Dewey, Ph.D., Barbara Gandek, M.S. How to score & interpret single item health status measures. Manual for users of SF8, Lincdn, RI. Quality Metric Incorporated, 2001. 1998-2001
- [Result] 1. ImmuKnow®® Cylex™ Immune Cell Function Assay, Package Insert (http://www.cylex.net/pdf/ImmuKnow_Insert-cx.pdf)